CLINICAL TRIAL: NCT06997029
Title: A Phase 1 First-in-human Study of BMS-986500 as Monotherapy in Advanced Solid Tumors and as Combination Therapy in CDK4/6 Inhibitor Pre-treated Advanced Breast Cancer
Brief Title: A Phase 1 Study of BMS-986500 as Monotherapy or Combination Therapy in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA243-0001; 2025-524334-26-00 (Other: EU CTR); U1111-1330-3304 (Other: WHO)
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumor; Advanced Breast Cancer; Advanced Ovarian Cancer
Keywords: cancer; oncology; solid tumor
MeSH Terms: conditions — Neoplasms | interventions — palbociclib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1A Monotherapy Dose Escalation (Experimental)
  Interventions: Drug: BMS-986500
- Part 1B Combination Dose Escalation (Experimental)
  Interventions: Drug: BMS-986500; Drug: Palbociclib; Drug: Fulvestrant
- Part 1C Monotherapy Pharmacodynamic (PD) Sub-study (Experimental)
  Interventions: Drug: BMS-986500
- Part 2A Monotherapy Dose Expansion (Experimental)
  Interventions: Drug: BMS-986500
- Part 2B Combination Dose Expansion (Experimental)
  Interventions: Drug: BMS-986500; Drug: Palbociclib; Drug: Fulvestrant

INTERVENTIONS:
Drug: BMS-986500 — Specified dose of specified days
Drug: Palbociclib — Specified dose on specified days
  Other Names: IBRANCE®; PD 0332991
  Arms: Part 1B Combination Dose Escalation; Part 2B Combination Dose Expansion
Drug: Fulvestrant — Specified dose on specified days
  Other Names: FASLODEX®
  Arms: Part 1B Combination Dose Escalation; Part 2B Combination Dose Expansion

SUMMARY:
The purpose of this study is to assess BMS-986500 as monotherapy in advanced solid tumors and as combination therapy in CDK4/6 inhibitor pre-treated advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥ 18 years of age.
* Participants must have histologically confirmed diagnosis of a locally advanced, unresectable, or metastatic solid tumor malignancy.
* Participants must have a measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Participants must have a stable Eastern Cooperative Oncology Group Performance Status of 0 or 1.
* For Part 2A only, participants must have CCNE1-amplified ovarian cancer

Exclusion Criteria:

* Participants must not have an active brain metastasis.
* Participants must not have impaired cardiac function or clinically significant cardiac disease.
* Participants must not have bleeding disorder or any history of clinically significant bleeding within the prior 3 months.
* Participants must not have Grade ≥ 2 peripheral neuropathy.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-12-14 (Estimated); Study Completion 2028-12-14 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Dose Limiting Toxicities (DLTs) | Up to Day 28 From Last Dose
Number of Participants With Adverse Events (AEs) | Up to Day 28 From Last Dose
Number of Participants With Serious Adverse Events (SAEs) | Up to Day 28 From Last Dose
Number of Participants With AEs Leading to Discontinuation | Up to Day 28 From Last Dose
Number of Participants With TEAEs Leading to Death | Up to Day 28 From Last Dose

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of BMS-986500 | Up to Approximately 2 Years
Time of Maximum Observed Serum Concentration (Tmax) of BMS-986500 | Up to Approximately 2 Years
Area Under the Concentration-time Curve Within a Dosing Interval (AUC(TAU)) of BMS-986500 | Up to Approximately 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (21):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Providence St. Jude Medical Center, Fullerton, California
  - Marin Cancer Care, Greenbrae, California
  - Moores Cancer Center, La Jolla, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Local Institution - 0008, Aurora, Colorado
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Local Institution - 0002, Lebanon, New Hampshire
  - Local Institution - 0014, Buffalo, New York
  - Northwell Health-Cancer Institute, New Hyde Park, New York
  - Local Institution - 0011, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - START Dallas Fort Worth, Fort Worth, Texas
  - NEXT Oncology, San Antonio, Texas
- Denmark (2):
  - Local Institution - 0024, Odense, Region Syddanmark
  - Local Institution - 0025, Copenhagen
- Japan (4):
  - Local Institution - 0021, Kashiwa, Chiba
  - Kansai Medical University Hospital, Hirakata, Osaka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06997029.html